CLINICAL TRIAL: NCT04973020
Title: A Single-centre, Single-dose, Open-label and Self-control Study to Evaluate the Effect of Efavirenz on Pharmacokinetic of SHR6390 in Healthy Chinese Subjects
Brief Title: A Drug-drug Interaction Study of SHR6390 on Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR6390-I-111
Record Dates: First submitted 2021-07-11; First posted 2021-07-22 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: The study is a single-center, open, single-dose, self-controlled clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: SHR6390、efavirenz

INTERVENTIONS:
Drug: SHR6390、efavirenz — SHR6390 tablet single dose；Efavirenz single dose.

SUMMARY:
The study is a single-center, open, single-dose, self-controlled clinical trial. It is planned to enroll 20 healthy adult subjects.Subjects will take the SHR6390 on Day1 and Day22 , and from Day8 to Day26 take the efavirenz.

ELIGIBILITY:
Inclusion Criteria:

1. The subject can communicate well with the researcher, understand and comply with the requirements of this study, and understand and sign the informed consent;
2. Healthy subjects aged 18~45 (including 18 and 45 years old);
3. Male body weight ≥ 50kg, female body weight ≥ 45kg, body mass index (BMI) within the range of 19 ~ 26kg /m2 (including 19 and 26 kg/m2) (BMI= weight (kg)/height 2 (m2));
4. The subjects had no fertility plan, took effective contraceptive measures voluntarily, and could not donate sperm or eggs within 7 months after signing the informed consent form to the last medication; the serum HCG test of women with fertility must be negative before the study medication.

Exclusion Criteria:

1. Anyone who has suffered from any clinical serious disease such as the circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatry and metabolic abnormalities, or any other disease which can affect the study results.
2. Those who have undergone surgery within 6 months before the trial, or plan to perform surgery during the study period;
3. Those who donated blood or suffered heavy blood loss (≥400 mL), received blood transfusions, or used blood products within 3 months before enrollment;
4. Have a history of allergies to drugs, food or other substances;
5. Those who have used soft drugs (such as marijuana) within 3 months before the test or hard drugs (such as cocaine, phencyclidine, etc.) within 1 year before the test; Those with positive results in urine drug abuse screening;
6. Those who have participated in any clinical trials and have taken study drugs within 3 months before the first administration;
7. Those who have taken any medicine within 4 weeks before the first administration (including prescription medicines, non-prescription medicines, Chinese herbal medicines, vitamins, calcium tablets and other food supplements), especially the drugs which have any effect on CYP3A4;
8. Regular drinkers within 6 months before the test, that is, drinking more than 14 units of alcohol per week (1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine), and any alcohol-containing products cannot be stopped during the study Those who are positive for alcohol breath test;
9. Those with any abnormal result (clinically significant) of vital signs, physical examination, 12-lead electrocardiogram, chest radiograph, abdominal ultrasound, colour Doppler echocardiography, hematology, clinical chemistry, urinalysis and coagulation;
10. Hepatitis B virus surface antigen is positive, or hepatitis C virus antibody is positive, or treponema pallidum antibody is positive, or human immunodeficiency virus antibody is positive.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Tmax | from Day 1 to Day 7 after the first dose and from Day 22 to Day 27 after the second dose
  Time to maximum observed serum concentration (Tmax) for SHR6390 after Single dose.
Cmax | from Day 1 to Day 7 after the first dose and from Day 22 to Day 27 after the second dose
  Maximum observed serum concentration (Cmax)for SHR6390 after Single dose.
AUC0-t | from Day 1 to Day 7 after the first dose and from Day 22 to Day 27 after the second dose
  Area under the plasma concentration versus time curve (AUC0-t) for SHR6390 after Single dose.
AUC0-inf | from Day 1 to Day 7 after the first dose and from Day 22 to Day 27 after the second dose
  Area under the plasma concentration versus time curve (AUC0-inf ) for SHR6390 after Single dose.
T1/2 | from Day 1 to Day 7 after the first dose and from Day 22 to Day 27 after the second dose
  Time to elimination half-life (T1/2) for for SHR6390 after Single dose.

SECONDARY OUTCOMES:
Number of subjects with adverse events and severity of adverse events | from Day 1 to Day 34 after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Beijing, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang J, Hu C, Zhang L. Effect of Efavirenz on the Pharmacokinetics of SHR6390 in Healthy Volunteers. Drug Des Devel Ther. 2024 Jul 19;18:3113-3119. doi: 10.2147/DDDT.S468478. eCollection 2024. PMID 39050802